CLINICAL TRIAL: NCT07183020
Title: Prospective, Multicentric, Real-world Investigation of Kappa Free Light Chains (KFLC) in Multiple Sclerosis (MS) and Clinically Isolated Syndrome (CIS)
Brief Title: Kappa Free Light Chains (KFLC) in Multiple Sclerosis (MS) and Clinically Isolated Syndrome (CIS)
Acronym: PRO-KFLC
Status: Enrolling by invitation | Type: Observational
Sponsor: Skripuletz, Thomas Prof. Dr. (Other)
Responsible Party: Sponsor-Investigator, Skripuletz, Thomas Prof. Dr., Prof. Dr. med., MD, Hannover Medical School
Organization: Hannover Medical School (Other)
Other Study IDs: 10167_B0_K2022
Record Dates: First submitted 2025-09-10; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome (CIS)
Keywords: multiple sclerosis; clinically isolated syndrome; cerebrospinal fluid; kappa free light chains; oligoclonal bands; biomarker; diagnosis
MeSH Terms: conditions — Multiple Sclerosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paired samples of serum and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis (MS) / clinically isolated syndrome (CIS): Patients diagnosed with multiple sclerosis (MS) or clinically isolated syndrome (CIS) and an available pair of cerebrospinal fluid (CSF) and serum
  Interventions: Diagnostic Test: Oligoclonal bands and kappa free light chains (KFLC)

INTERVENTIONS:
Diagnostic Test: Oligoclonal bands and kappa free light chains (KFLC) — Comparison of oligoclonal bands and kappa free light chains (KFLC) in patients with multiple sclerosis (MS) / clinically isolated syndrome (CIS)

SUMMARY:
The goal of this observational study is to learn about the role of kappa free light chains (KFLC) in cerebrospinal fluid (CSF) in the diagnosis of multiple sclerosis (MS) and clinically isolated syndrome (CIS). The main question it aims to answer is:

Are KFLC superior, inferior or equally useful in the diagnostic work-up of CSF of patients with MS and CIS?

In CSF and serum sample pairs of patients diagnosed with MS or CIS, KFLC are measured using a nephelometric assay and are compared with the gold standard, of CSF diagnostics, oligoclonal bands.

DETAILED DESCRIPTION:
In this multicenter study, paired cerebrospinal fluid (CSF) and serum samples from patients with chronic inflammatory diseases of the central nervous system (multiple sclerosis (MS) / clinically isolated syndrome (CIS)) are investigated to evaluate the diagnostic utility of CSF-specific oligoclonal bands and kappa free light chains (KFLC). Both biomarkers have already demonstrated diagnostic relevance in this patient population, but comparative multicenter studies are still lacking. Another key challenge for the clinical implementation of KFLC is the absence of standardized reference values, as different cut-offs were proposed.

To address this gap, CSF-specific oligoclonal bands and KFLC are prospectively analyzed in a multicenter cohort of patients with MS / CIS. Samples and associated data are collected prospectively and partially retrospectively from participating centers. Included patients are followed longitudinally to determine whether conversion from CIS to clinical definite MS occurs and to monitor disease progression over time.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with multiple sclerosis (MS) or clinically isolated syndrome (CIS) according to 2017-revised McDonald criteria for MS
* age between 18 and 70 years

Exclusion Criteria:

* no diagnosis of MS or CIS according to 2017-revised McDonald criteria for MS
* no available cerebrospinal fluid (CSF) and serum sample pairs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being adult, diagnosed with multiple sclerosis (MS) or clinically isolated syndrome (CIS), receiving a cerebrospinal fluid (CSF) analysis as part of the clinical routine diagnostic work-up
Sampling Method: Non-Probability Sample
Enrollment: 1142 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of diagnostic sensitivity of cerebrospinal fluid (CSF) kappa free light chains (KFLC) in multiple sclerosis (MS) and clinically isolated syndrome (CIS) compared to oligoclonal bands | From study inclusion to the final analysis of cerebrospinal fluid (CSF) oligoclonal bands and kappa free light chains (KFLC) at 12 months
  Evidence of an intrathecal kappa free light chains (KFLC) synthesis is equally sensitive to assess for an intrathecal immunglobulin synthesis compared with oligoclonal bands

SECONDARY OUTCOMES:
Superiority of Reiber´s diagram for kappa free light chains (KFLC) compared to KFLC index of 6.1 to assess for an intrathecal KFLC synthesis in multiple sclerosis (MS) and clinically isolated syndrome (CIS) patients | From study inclusion to the final analysis of cerebrospinal fluid (CSF) oligoclonal bands and kappa free light chains (KFLC) at 12 months
  The frequence of an intrathecal kappa free light chains (KFLC) synthesis as assessed by Reiber´s diagram is significantly higher as compared to the KFLC index of 6.1 as cut-off

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Hochschule Hannover / Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Pseudonym, immunoglobulin (Ig) G serum (g/l), IgG cerebrospinal fluid (CSF) (mg/l), Q IgG, Albumin serum (g/l), Albumin CSF (mg/l), Q-Albumin
Time Frame: 27.10.2022 beginning ending 10 years after publication
Access Criteria: Individual participant data (IPD) will be stored and processed in pseudonymized form on the server of the computing center of Hannover Medical School (MHH) in compliance with data protection regulations, in particular the EU General Data Protection Regulation (GDPR). Access to the pseudonymized data and their processing will be restricted to authorized study team members who are bound by confidentiality obligations. Unused data will be deleted. Remaining data will be archived for ten years after study completion in accordance with good scientific practice guidelines and will be irreversibly deleted thereafter. No external parties will have access to the IPD or supporting information.

REFERENCES:
- [Background] Schwenkenbecher P, Konen FF, Wurster U, Jendretzky KF, Gingele S, Suhs KW, Pul R, Witte T, Stangel M, Skripuletz T. The Persisting Significance of Oligoclonal Bands in the Dawning Era of Kappa Free Light Chains for the Diagnosis of Multiple Sclerosis. Int J Mol Sci. 2018 Nov 29;19(12):3796. doi: 10.3390/ijms19123796. PMID 30501024
- [Background] Schwenkenbecher P, Konen FF, Wurster U, Witte T, Gingele S, Suhs KW, Stangel M, Skripuletz T. Reiber's Diagram for Kappa Free Light Chains: The New Standard for Assessing Intrathecal Synthesis? Diagnostics (Basel). 2019 Nov 16;9(4):194. doi: 10.3390/diagnostics9040194. PMID 31744096
- [Background] Konen FF, Wurster U, Witte T, Jendretzky KF, Gingele S, Tumani H, Suhs KW, Stangel M, Schwenkenbecher P, Skripuletz T. The Impact of Immunomodulatory Treatment on Kappa Free Light Chains as Biomarker in Neuroinflammation. Cells. 2020 Mar 31;9(4):842. doi: 10.3390/cells9040842. PMID 32244362
- [Background] Konen FF, Schwenkenbecher P, Jendretzky KF, Gingele S, Suhs KW, Tumani H, Susse M, Skripuletz T. The Increasing Role of Kappa Free Light Chains in the Diagnosis of Multiple Sclerosis. Cells. 2021 Nov 6;10(11):3056. doi: 10.3390/cells10113056. PMID 34831279
- [Background] Susse M, Konen FF, Schwenkenbecher P, Budde K, Nauck M, Grothe M, Hannich MJ, Skripuletz T. Decreased Intrathecal Concentrations of Free Light Chains Kappa in Multiple Sclerosis Patients Taking Very High Effective Disease-Modifying Treatment. Diagnostics (Basel). 2022 Mar 16;12(3):720. doi: 10.3390/diagnostics12030720. PMID 35328273
- [Background] Konen FF, Schwenkenbecher P, Jendretzky KF, Gingele S, Witte T, Suhs KW, Grothe M, Hannich MJ, Susse M, Skripuletz T. Kappa Free Light Chains in Cerebrospinal Fluid in Inflammatory and Non-Inflammatory Neurological Diseases. Brain Sci. 2022 Apr 3;12(4):475. doi: 10.3390/brainsci12040475. PMID 35448006
- [Background] Konen FF, Hannich MJ, Schwenkenbecher P, Grothe M, Gag K, Jendretzky KF, Gingele S, Suhs KW, Witte T, Skripuletz T, Susse M. Diagnostic Cerebrospinal Fluid Biomarker in Early and Late Onset Multiple Sclerosis. Biomedicines. 2022 Jul 7;10(7):1629. doi: 10.3390/biomedicines10071629. PMID 35884934
- [Background] Hannich MJ, Konen FF, Gag K, Alkhayer A, Turker SN, Budde K, Nauck M, Wurster U, Dressel A, Skripuletz T, Susse M. Implications of monoclonal gammopathy and isoelectric focusing pattern 5 on the free light chain kappa diagnostics in cerebrospinal fluid. Clin Chem Lab Med. 2024 Jul 23;63(1):147-153. doi: 10.1515/cclm-2023-1468. Print 2025 Jan 29. PMID 39039726
- [Background] Konen FF, Wurster U, Schwenkenbecher P, Gerritzen A, Gross CC, Eichhorn P, Harrer A, Isenmann S, Lewczuk P, Lewerenz J, Leypoldt F, Otto M, Regeniter A, Roskos M, Ruprecht K, Spreer A, Strik H, Uhr M, Wick M, Wildemann B, Wiltfang J, Zimmermann T, Hannich M, Khalil M, Tumani H, Susse M, Skripuletz T; German Society for Cerebrospinal Fluid Diagnostics and Clinical Neurochemistry (DGLN e.V.). Oligoclonal bands and kappa free light chains: Competing parameters or complementary biomarkers? Autoimmun Rev. 2025 Apr 30;24(5):103765. doi: 10.1016/j.autrev.2025.103765. Epub 2025 Feb 11. PMID 39947571